CLINICAL TRIAL: NCT06803966
Title: Comparison of Rescue Analgesia Requirement After Transversus Abdominal Plane (TAP) Block Vs Local Anesthetic Wound Infiltration After Laparoscopic Cholecystectomy
Brief Title: Comparison of Rescue Analgesia Requirement in Patients Undergoing Laparoscopic Cholecystectomy After Transversus Abdominal Plane (tap) Block Vs Local Anesthetic Wound Infiltration At the End of Surgery
Acronym: TAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fazaia Ruth Pfau Medical College (Other)
Responsible Party: Principal Investigator, Sumbul Andleeb, Principal Investigator, Fazaia Ruth Pfau Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FazaiaRuthPfauMC
Record Dates: First submitted 2025-01-22; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Rescue Analgesia
Keywords: transversus abdominal plane block; local anesthetic wound infiltration

STUDY DESIGN:
Intervention Model Description: group A will get local ansthetic wound infiltration at port site and Group b will get Transversus abdominal plane block
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: local anesthetic infiltration at port sites (Active Comparator): Group A patient's will receive local anesthetic wound infiltration at port sites with inj Bupivacaine (Bupivacaine Hydrochloride) 0.5%
  Interventions: Other: Post Operative Analgesia
- Group B : TAP block (Active Comparator): Group b will receive Transversus Abdominal Plane (TAP) block at both sides using inj bupivacaine (Bupivacaine Hydrochloride) 0.25%
  Interventions: Other: Post Operative Analgesia

INTERVENTIONS:
Other: Post Operative Analgesia — Group A will receive local wound infiltration at port sites with inj bupivacaine (bupivacaine Hydrochloride) 0.5 %
  Group B will receive Transversus Abdominal Plane Block on both sides by inj bupivacaine (bupivacaine Hydrochloride) 0.25%
  Other Names: Group A : local wound infiltration; Group B : TAP block

SUMMARY:
patients undergoing laparoscopic cholecystectomy will be diveided into 2 groups A & B . Group A will receive local anesthetic wound infiltration and group B will receive Transversus abdominal plane block as a post operative analgesia. the time for request of first rescue analgesia between the 2 groups will be compared

DETAILED DESCRIPTION:
After acquiring approval from Institutional Review Board, the work on the study will begin. The patients planned to undergo elective laparoscopic cholecystectomy first appear for pre-anesthesia assessment and here all relevant baseline tests and demographics (age, weight, ASA score, co morbid and allergies) will be recorded. The patient meeting the inclusion criteria will be explained about the study in the language they understand, its benefits, risks and any other relevant queries will be heard and answered. Those willing to participate will be enrolled into the study, after written consent. Confidentiality of the study subjects will be assured throughout. Data will only be accessible to the principal investigator.

Patients will be assigned either in Group A or Group B using sequentially numbered opaque sealed envelope protocol. Both patients and study investigators will be blinded to study groups. Only an anesthetist who will prepare the medication and will not be part of this study, will have correct knowledge of group identification.

On the day of operation, after patient is shifted to the operating room, monitors will be attached and vitals including Blood pressure, heart rate, mean arterial blood pressure, SpO2 and ETCO2 will be continuously monitored. Patient will be pre medicated by 0.1 mg/kg nalbuphine. For induction of anesthesia, 2 mg/kg propofol and 0.5 mg/kg Atracurium as a relaxant will be given. Anesthesia will be maintained on Isoflurane. Before the start of procedure NG tube will be inserted.

At the end of surgery before extubating, Injection ondansetron 0.15 mg/kg IV will be given to the patient. Next, as patients will be divided into two groups via closed envelope method, Group A will get local anesthetic wound infiltration and group B will receive TAP block. Local Anesthetic infiltration will be given with 20ml of 0.5% bupivacaine (5ml at each port site). TAP block will be given as 0.25% bupivacaine 20ml on each side, using ultrasound guidance.

After extubation, patient will be shifted to post surgical ward where they will be kept under close monitoring. Pain status will be monitored using the NRS at following hours 0, 2, 4, 8, 12, 24 and/or when patient complains. Rescue analgesia will be given by injection Toradol as 30 mg IV, when patient categorizes the pain as 4 or more according to NRS. This time at which rescue analgesia is given will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* both gender patients undergoing elective laparoscopic cholecystectomy ASA physical status classification 1 & 2

Exclusion Criteria:

* patients with chronic pain patients unable to understand NRS pain scale conversion of laparoscopic to open cholecystectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-01-11 (Actual)

PRIMARY OUTCOMES:
first rescue analgesia | from enrollment to 24 hours post operation
  time of requirement of first rescue analgesia will be compared between group a and group b

CONTACTS AND LOCATIONS:
Locations (1):
- PAF hospital Faisal base, Karachi, Sindh, Pakistan